CLINICAL TRIAL: NCT04139863
Title: Pilot Study on Oral Health Status Chairside Mouthrinse Test in Finnish Adolescents and Cost Effectiveness of the Test
Brief Title: Chairside Mouthrinse Test and Cost Effectiveness
Acronym: JuvePar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Teija Raivisto, Principal Investigator, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JuvePar
Record Dates: First submitted 2019-10-07; First posted 2019-10-25 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Periodontitis, Juvenile
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aMMP-8 chairside test (Other): Test group. The aMMP-8 chairside mouth rinse test is performed for the test group.It identifies adolescents with poor oral hygiene at risk for subclinical periodontitis without detectable and visible manifestations of the illness, such as periodontal deepened pockets.
  Interventions: Diagnostic Test: aMMP-8 chairside test
- No test (No Intervention): The other group is control group. No test administered.

INTERVENTIONS:
Diagnostic Test: aMMP-8 chairside test — No test
  Other Names: No test
  Arms: aMMP-8 chairside test

SUMMARY:
The aim is to study whether participants at risk could be identified using an aMMP-8 chairside mouth rinse test and to study if oral health and health behaviour is linked to the test result in Finnish adolescents.

DETAILED DESCRIPTION:
Adolescents (14-15-year-olds) are randomly divided to control group and test group. Chairside mouth rinse test for aMMP-8 is performed for the test group. Two groups are compared with each other.

Participants are asked to fill a questionnaire which consists of questions concerning oral hygiene habits, tobacco products, alcohol, drug and snuff use.

ELIGIBILITY:
Inclusion Criteria:

* All 8 class (aged 14-15 years) pupils in Jukola, Hämeenlinna, Finland
* Written informed consent from the participants and their parents (one of them)

Exclusion Criteria:

* No written consent to the study

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-11-02 (Estimated); Study Completion 2020-11-02 (Estimated)

PRIMARY OUTCOMES:
aMMP-8 test | 1 year
  Mouth rinse samples are analysed by method for chair-side diagnostic testing: the aMMP-8 specific lateral-ﬂow point-of-care (PoC)/chair-side test (PerioSafe®, Dentognostics GmbH, Jena, Germany). The result is provided in 5 minutes and is graded by eye as positive or negative. One line means that the test is negative but successfully done and two lines the test is positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Maria Heikkinen, Helsinki, Helsinki University, Finland

IPD SHARING:
Plan to Share IPD: No